CLINICAL TRIAL: NCT01114022
Title: Comparison of Prevention Bacterial Inhalation of Patients on Mechanical Ventilation by Using Endotracheal Tube Balloon Polyvinyl Chloride or Polyurethane
Brief Title: Prevention Inhalation of Bacterial by Using Endotracheal Tube Balloon Polyvinyl Chloride or Polyurethane
Acronym: Top-cuff
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Kimberly-Clark Corporation (Industry); Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OST08029; ID RCB2008 -A007 12-53 (Registry Identifier: AFSSAPS)
Record Dates: First submitted 2010-04-29; First posted 2010-04-30 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Acute Respiratory Failure; Mechanical Ventilation Complication
Keywords: Acute respiratory failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Active comparator (Active Comparator): cylindrical PVC cuff
  Interventions: Device: Active comparator
- Experimental 1 (Experimental): cylindrical polyurethane cuff
  Interventions: Device: Experimental 1
- Experimental 2 (Experimental): conic PVC cuff
  Interventions: Device: Experimental
- Experimental 3 (Experimental): conic polyurethane cuff
  Interventions: Device: experimental 3

INTERVENTIONS:
Device: Experimental 1 — oeso pharyngeal device
  Other Names: oeso pharyngeal device
  Arms: Experimental 1
Device: Experimental — oeso pharyngeal device
  Other Names: oeso pharyngeal device
  Arms: Experimental 2
Device: experimental 3 — oeso pharyngeal device
  Other Names: oeso pharyngeal device
  Arms: Experimental 3
Device: Active comparator — oeso pharyngeal device
  Other Names: oeso pharyngeal device
  Arms: Active comparator

SUMMARY:
A number of techniques have been recommended for the prevention of ventilator acquired pneumonia (VAP). These techniques - such as patient positioning, continuous sub-glottic suction of the secretions, selective decontamination of the digestive tract etc… - aim at prevent the inhalation of oro-pharyngeal contaminated secretions around the cuff of the tracheal tube used for connecting the patient to the machine. Their efficacy has been regularly challenged and they are still unable to suppress totally the occurrence of VAP. The cuff of the tracheal tube used for long-term MV in the ICU is most often a low pressure high volume polyvinyl chloride (PVC) cuff in order to adhere to a large surface of the tracheal wall without inducing ischemic lesions. Recent advances allowed industrial companies to provide us with 1) polyurethane cuffs and 2) cuffs with a conic shape, both potentially offering a better tightness against inhalation at least in VITRO and in animal models. The effect on the reduction of VAP incidence has been suggested by several pilot series. The aim of the present project is to assess the efficacy of four types of cuffs (PVC with a conic or a cylinder shape and polyurethane with a conic or a cylinder shape) to prevent tracheal colonisation. We shall measure both oro-pharyngeal and tracheal colonisation during the hours and days following intubation. This will be done in 600 ICU patients of four university affiliated centres from France and Tunisia divided in 64 cluster randomized groups. The results of this research will confirm (or not) the rationale to perform a larger study designed specifically to address the impact on VAP.

DETAILED DESCRIPTION:
Long-term mechanical ventilation (MV) is a risk factor for acquisition of bacterial pneumonia because the tracheal tube by-passes the natural mechanisms of airway protection, and particularly epiglottis and trachea-bronchial mucosa. Acute respiratory failure and potential associated organ dysfunctions require that MV patients are sedated and sometimes in strict horizontal supine position. Sedation and conscience alteration do not permit to swallow oro-pharyngeal secretions, and horizontal position favors bacterial colonization and secretions stagnation in the posterior part of the pharynx. These aspects favor iterative inhalation of oro-pharyngeal secretions around the cuff of the tracheal tube. The cuff, which principal objective is to permit the pressurization of lower respiratory tract during the inspiratory phase by preventing air leak around the tracheal tube, allows a certain degree of protection of the tracheal tree against micro-inhalations. Using diagnostic criteria of Ventilator associated pneumonia (VAP) based on distal protected samples, their incidence is around 10 per 1,000 MV-days in medical-surgical ICUs. These VAP are associated to an attributable mortality around 25%. A number of recommendations have been established to prevent VAP occurrence. The 45° semi-recumbent positioning of the patient 's reduces gastro-esophageal reflux and VAP incidence. This result is limited by the fact that a 45° inclination is not routinely obtained in every patients (30° would not give the same result ) and that several studies have shown conflicting results. The continuous suction of the secretions above the cuff is very logical but its efficacy has been challenged, partly because technical failures due to the occlusion of the aspiration system and because gravity prevents the tracheal secretions clearance. The selective decontamination of the digestive tract is effective particularly to prevent early VAP, but is limited by its potential role in the global increase in resistance to antibiotics. Oral decontamination with Chlorhexidine or iodine polyvidon reduce VAP. Using drugs which increases the gastric pH to prevent stress ulcers favors gastric bacterial growth and VAP. Using gastric pro-kinetics or post-pyloric enteral nutrition do not reduce VAP. Alternate prone positioning, has not been proven to improve the outcome of ARDS patients but reduces the incidence of VAP, potentially because it favors pharyngeal drainage through the mouth. The use of heat and moisture exchangers to limit airways drying with ventilation, seems better than heat humidifiers to reduce VAP. Recently, the use of an positive end expiratory pressure (PEEP) was shown to reduce the volume on inhalations around the cuff. Finally, mask ventilation, by preserving upper airways integrity, in those cases it allows a sufficient ventilation replacement, is associated to a substantial reduction in VAP.

In those patients ventilated through an oro-tracheal tube, the rational use of the above mentioned techniques allows to reach a low VAP incidence rate, but not to completely eradicate these infections.

The cuffs of the tracheal tubes which are currently recommended and routinely used in long-term (more than 2 days) ventilation are made of polyvinyl chloride and have a high volume cylindrical shape, allowing a low pressure after inflation, designed to cover the tracheal wall without inducing ischemic lesions of the tracheal mucosa. Such lesions are responsible for laryngeal edema - a clinical stridor after extubation occurs in around 12% of patients -, and rarely for granuloma and stenosis which induce sequelae which are disabling and/or difficult to repair with surgery. The use of tube coated with antiseptics is currently under investigation. Protection against tracheal lesions induced by the tracheal tube requires a regular and frequent assessment of the cuff pressure over the day and night time. Recent experimental studies showed that these cuffs are bad protectors against micro-inhalations around the cuff. Several companies provide us with new polyurethane cuff tubes, which physical characteristics are associated - in VITRO, on animal tracheas, and during general anesthesia to a better tightness than polyvinyl chloride cuffs. They also provide us with conic shaped cuffs, made out of either PVC or polyurethane. Authors found that the Hi-Lo and the SEALGUARD cuffs have similar capabilities to prevent against methylene blue leakage, and others did not find a preventive effect of the pressure control of the Hi-Lo cuff against VAP. A reduction of early VAP was observed in one series after cardiac surgery.

Our hypothesis is that the tracheal tubes with a polyurethane and/or a conic shaped cuff are associated with a lower colonization of the tracheal tree during the days following tracheal intubation, than tubes with a cylindrical polyvinyl chloride cuff. The patients will be allocated to randomized clusters into four groups : 1) cylindrical PVC cuff, 2) cylindrical polyurethane cuff, 3) conic PVC cuff and 4) conic polyurethane cuff. In the four groups, the tubes will be inserted with the conventional technique of tracheal intubation under general anesthesia and direct laryngoscopy, inside the ICU. The tube cuff will be immediately inflated to a 25 cm of water or at the plateau pressure level of the ventilator in case it is higher than 25 cm of water according to the current recommendations. The tracheal tube will be connected to the ventilator, set in a volume or pressure control mode with a minimal PEEP of 5 cm of water.

The research will be conducted according to the protocol, following the good clinical practices and current recommendations about MV and Intensive Care practices proposed by the French Society of Intensive Care Medicine (www.srlf.org) and the European Society of Intensive Care Medicine (www.ESICM.org).

Principal endpoint(s) : quantitative assessment of bacterial colonization in the oro-pharyngeal (above the cuff) and tracheal (below the cuff) secretions at 2 hours (H2), 1 day (D1), D2 and D3 after intubation. The collection of the secretions above and below the cuff will allow to document the origin of the tracheal bacteria. The bacterial quantity at each sampling will be compared between the patients groups to establish the role of the cuff in the antibacterial protection of the lower airway.

The oro-pharyngeal and tracheal samples will be performed 2 hours after oro-pharyngeal application of Chlorhexidine and a tracheal aspiration. Bacterial cultures will be done on standard media and the quantitative cultures will be carried out by serial dilution of the samples.

Secondary endpoints :

VAP occurrence : the diagnosis of VAP will be based on the positive results of a protected specimen brush (over 103 cfu/mL) or a broncho-alveolar lavage (over 2 % infected cells or over 104 cfu/mL). Distal bronchial samples will be performed under fiberoptic bronchoscopy when several of the following criteria suggestive VAP will be present, corresponding to a CPIS score at least equal to 6 : fever, new chest X-ray opacity, hyper-leucocytosis, arterial oxygenation alteration.

Cross-over cluster randomization : an individual randomization is almost impossible to achieve, because of the emergency setting of any decision of tracheal intubation in the ICU. Therefore we chose to ascribe random periods during which every tracheal tubes of the ICU will be those of the study protocol for the given period. The random plan will be different in each participating ICU. Each ICU will have to perform periods of 10 patients. Each ICU intend to recruit 10 patients in periods of around 2 months. The physicians in charge of the patients will be kept blind of the bacteriological samples results. This will prevent them to modify their clinical practices according to these results and particularly to influence their clinical suspicion of VAP and/or stridor.

ELIGIBILITY:
Inclusion criteria :

* patients which duration of tracheal intubation expected by the physician is more than 24 h
* patients intubated by one of the participating ICU
* adult patients (> 18 years).

Exclusion criteria :

* Recent (less than a month) tracheal or bronchial surgery.
* Bronchial dilation or cystic fibrosis
* Non-intubated patients in ICUs or emergency rooms participating centers.
* Intubation> 24 hours in the previous 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620 (Actual)
Dates: Start 2010-09; Primary Completion 2014-03 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Whether the probes tracheal intubation with a polyurethane balloon or balloon-shaped tapered, or both at once, due to their better seal, are associated with reduced colonization routes from bronchial secretions oro-pharynx | 7 days

SECONDARY OUTCOMES:
To determine the impact of PAVM | one month
To determine the incidence of laryngeal dyspnea with each probe | one month

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Misset, MD PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Groupe Hospitalier St Joseph, Paris, France

REFERENCES:
- [Background] Misset B, Timsit JF, Dumay MF, Garrouste M, Chalfine A, Flouriot I, Goldstein F, Carlet J. A continuous quality-improvement program reduces nosocomial infection rates in the ICU. Intensive Care Med. 2004 Mar;30(3):395-400. doi: 10.1007/s00134-003-2096-1. Epub 2003 Dec 12. PMID 14673521
- [Background] Koenig SM, Truwit JD. Ventilator-associated pneumonia: diagnosis, treatment, and prevention. Clin Microbiol Rev. 2006 Oct;19(4):637-57. doi: 10.1128/CMR.00051-05. PMID 17041138
- [Background] Garrouste-Orgeas M, Chevret S, Arlet G, Marie O, Rouveau M, Popoff N, Schlemmer B. Oropharyngeal or gastric colonization and nosocomial pneumonia in adult intensive care unit patients. A prospective study based on genomic DNA analysis. Am J Respir Crit Care Med. 1997 Nov;156(5):1647-55. doi: 10.1164/ajrccm.156.5.96-04076. PMID 9372689
- [Background] Dullenkopf A, Schmitz A, Frei M, Gerber AC, Weiss M. Air leakage around endotracheal tube cuffs. Eur J Anaesthesiol. 2004 Jun;21(6):448-53. doi: 10.1017/s0265021504006064. PMID 15248624
- [Background] Lucangelo U, Zin WA, Antonaglia V, Petrucci L, Viviani M, Buscema G, Borelli M, Berlot G. Effect of positive expiratory pressure and type of tracheal cuff on the incidence of aspiration in mechanically ventilated patients in an intensive care unit. Crit Care Med. 2008 Feb;36(2):409-13. doi: 10.1097/01.CCM.0000297888.82492.31. PMID 18007268
- [Derived] Philippart F, Gaudry S, Quinquis L, Lau N, Ouanes I, Touati S, Nguyen JC, Branger C, Faibis F, Mastouri M, Forceville X, Abroug F, Ricard JD, Grabar S, Misset B; TOP-Cuff Study Group. Randomized intubation with polyurethane or conical cuffs to prevent pneumonia in ventilated patients. Am J Respir Crit Care Med. 2015 Mar 15;191(6):637-45. doi: 10.1164/rccm.201408-1398OC. PMID 25584431